CLINICAL TRIAL: NCT05348889
Title: A Phase 1/2, First in Human, Single-arm, Open-label Study to Evaluate the Safety and Efficacy of Triple-specific T-cell Engager 1A46 in Adult Patients with Advanced CD20 And/or CD19 Positive B-cell Hematologic Malignancies
Brief Title: First-in-Human (FIH) Trial of 1A46 in Subjects with Advanced CD20 And/or CD19 Positive B-cell Hematologic Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's Research and Development strategy adjustment
Sponsor: Chimagen Biosciences, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG1A46-US01
Record Dates: First submitted 2022-03-29; First posted 2022-04-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Non-Hodgkin's Lymphoma (disorder); Acute Lymphoid Leukemia, Disease (disorder)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Experimental): Open label, single arm trial where 1A46 will be administered
  Interventions: Drug: 1A46 Injection

INTERVENTIONS:
Drug: 1A46 Injection — Participants will receive IV 1A46 weekly for Cycles 1-8, then every 3 weeks (Q3W) for Cycles 9-16 (21 days/cycle).
  Other Names: CMG1A46

SUMMARY:
This study will evaluate the safety and efficacy of 1A46 in adult patients with advanced CD20 and/or CD19 positive B-cell non-Hodgkin's lymphoma (NHL) or acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This study is an open-label, multicenter, 2-part study of 1A46 in adult patients with advanced relapsed/refractory (r/r) CD20 and/or CD19 positive B-cell non-Hodgkin lymphoma (NHL) and B-cell acute lymphoblastic leukemia (ALL) who do not have effective standard treatment available. This FIH study will include a dose escalation part and a dose expansion part in 4 cohorts.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Part:

Aggressive NHL Patients：

* Aggressive NHL including mantle cell lymphoma and DLBCL histologies, NOS and/or BCL2, BCL6, and or MY B-cell lymphoma with intermediate features between DLBCL, FL grade 3B, and aggressive B-cell lymphoma unclassifiable
* have previously R-CHOP, R-EPOCH or equivalent anti-CD20 containing therapy
* with ≥ 2 prior lines of systemic therapy
* received or ineligible for autologous stem cell transplant (ASCT)
* have received or been intolerant of all other standard therapies thought to confer clinical benefit.

Indolent NHL Patients:

* including FL of Grades 1-3A and marginal zone lymphoma (MZL)
* refractory or relapsed after ≥ 2 prior lines of systemic therapy who have received or been intolerant of all other standard therapies thought to confer clinical benefit.
* Patients must require systemic therapy based on disease-specific criteria.

NHL patients should meet the following requirements:

* The following considerations pertain to prior treatment regimens for NHL:

  1. Preinduction salvage chemotherapy and ASCT should be considered 1 therapy.
  2. Patients with gastric extranodal MZL, should have failed H. pylori eradication therapy (when H. pylori positive).
* NHL patients must have expression of CD20 and/or CD19-expression
* NHL patients in the dose escalation part of the study must have ≥ 1 measurable target lesion as defined by Lugano 2014 criteria ALL Patients：

Ph-positive or Ph-negative B-cell ALL refractory to or relapsed after frontline treatment and 1 salvage regimen, have received or been intolerant of all other standard therapies thought to confer clinical benefit. ALL patients should meet the following requirements:

* Relapsed after or not a candidate for allogeneic SCT.
* No active acute or chronic graft-versus-host disease for 2 months prior to enrollment and currently receiving no immunosuppressive therapy.
* persistent CD19 staining of ≥ 50% of blasts.

Exclusion Criteria:

* Patient has brain metastasis or other significant neurological conditions.
* Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period.
* Active serious infection requiring antibiotics within 14 days before study entry.
* Treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or immunosuppressive medication ≤ 7 days before the first dose of 1A46, with the following exceptions:

  1. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroids.
  2. Dexamethasone used to reduce peripheral blast counts in ALL patients.
* Active hepatitis B or C.
* Known human immunodeficiency virus (HIV) infection.
* Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.
* Cerebrovascular accident, transient ischemic attack, myocardial infarction, unstable angina, or New York Heart Association class III or IV heart failure < 6 months of study entry; uncontrolled arrhythmia < 3 months of study entry.
* Major surgery < 4 weeks or minor surgery < 2 weeks prior to screening.
* Live virus vaccines < 30 days prior to screening.
* Inflammatory chronic diseases, or any other diseases the investigator considers can be exacerbated in the setting of immune activation.
* History of Grade 3-4 allergic reaction to treatment with another mAb, or known to be allergic to protein drugs or recombinant proteins or excipients in 1A46 drug formulation.
* Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma in situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
* History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies.
* Pleural effusion, pericardial effusion or ascites requiring frequent drainage or medical intervention.
* QTc > 480 msec using Fredericia's QT correction formula
* Patients in the dose escalation part who weigh < 40 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Escalation: Incidence of Adverse Events | Adverse Events are assessed during the first cycle (28 days) in each cohort
  To assess the safety and tolerability of 1A46
Escalation: Dose liming toxicity (DLT) | DLTs are assessed during the first cycle (28 days) in each cohort
  To identify the RP2D and the MTD, if reached

SECONDARY OUTCOMES:
Escalation: Maximum observed concentration (Cmax) | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Time to reach Cmax (Tmax) | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Area Under the Concentration-Time Curve (AUC) from Time 0 to t | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Area under the serum concentration-time curve from time 0 to infinity (AUCinf) | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Terminal disposition phase half-life(t1/2) | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Total clearance after IV administration (CL) | At enrollment and at multiple timepoints until treatment discontinuation, assessed up to 1 year
  To characterize the PK properties of 1A46
Escalation: Anti-drug antibody (ADA) | From Baseline up to end of study or discontinuation due to disease progression, up to 5 years
  To characterize the PK properties of 1A46
Escalation: Objective Response Rate (ORR) | From Baseline up to end of study or discontinuation due to disease progression, up to 5 years
  To evaluate preliminary anti-tumor efficacy of 1A46
Escalation: Disease control rate (DCR) | From Baseline up to end of study or discontinuation due to disease progression, up to 5 years
  To evaluate preliminary anti-tumor efficacy of 1A46
Escalation: Progression free survival (PFS) | From Baseline up to end of study or discontinuation due to disease progression, up to 5 years
  To evaluate preliminary anti-tumor efficacy of 1A46
Escalation: Overall survival (OS) | From Baseline up to end of study or discontinuation due to disease progression, up to 5 years
  To evaluate preliminary anti-tumor efficacy of 1A46

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Chimagen Biosciences, Ltd
Locations (5):
- United States (5):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Norton Cancer Institute, Louisville, Kentucky
  - UPMC CancerCenter, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert & the Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No